CLINICAL TRIAL: NCT01366066
Title: Transcutaneous Mechanical Nerve Stimulation (TMNS) by Vibration in the Treatment of Stress Incontinence and Urge Incontinence
Brief Title: Transcutaneous Mechanical Nerve Stimulation in the Treatment of Incontinence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to recruit participants
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2010-109
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Stress Urinary Incontinence; Urge Urinary Incontinence
Keywords: Stress incontinence; urge incontinence; overactive bladder syndrome; vibration; nerve stimulation
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TMNS treatment - Stress incontinence (Active Comparator): Women with stress incontinence treated with active TMNS (vibration)
  Interventions: Device: Transcutaneous mechanical nerve stimulation
- No treatment - stress incontinence (No Intervention): Women with stress incontinence NOT treated with TMNS (vibration)
- TMNS treatment - Urge incontinence (Active Comparator): Women with stress incontinence treated with TMNS (vibration)
  Interventions: Device: Transcutaneous mechanical nerve stimulation
- No treatment - urge incontinence (No Intervention): Women with urge incontinence NOT treated with TMNS (vibration)

INTERVENTIONS:
Device: Transcutaneous mechanical nerve stimulation — A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Denmark) will be used. The stimulation works through a vibrating disc of hard plastic with a diameter of 3.5 cm. The stimulation point will be the perineum. The stimulation will be performed with a vibration amplitude of 2 mm and a frequency of 100 Hz.
  A daily stimulation sequence consisting of 10 seconds of stimulation followed by a 10 second pause repeated 10 times will be used through 6 weeks.
  Other Names: FERTI CARE personel, Multicept A/S, Albertslund, Danmark
  Arms: TMNS treatment - Stress incontinence; TMNS treatment - Urge incontinence

SUMMARY:
During transcutaneous mechanical nerve stimulation in spinal cord injured men an increase in pressure was observed in the external urethral sphincter along with an increase in bladder capacity. In a subsequent study it was demonstrated that Transcutaneous Mechanical Nerve Stimulation (TMNS) in women could induce pressure increment of the external urethral sphincter. A pilot study have since shown that after 6 weeks of stimulation 24 out of 33 women suffering from urinary stress incontinence were able to contract their pelvic floor muscles and had become free of symptoms. Another pilot study has shown promising effect on the overactive bladder syndrome.

The present study aims to treat urinary incontinence and includes 2 groups of patients with 30 patients in each group: Women suffering from urinary stress incontinence and women suffering from urge incontinence. A medical vibrator is used and in each group the subjects will be randomized to vibration treatment or no vibration treatment. All patients will receive pelvic floor training and all women suffering from urge incontinence will receive anticholinergic medications.

The stimulation will be performed at the perineum every day for 6 weeks with an amplitude of 2 mm and a frequency of 100 Hz. Results will be evaluated on the basis of questionnaires, micturition diaries and diaper tests.

If the investigators are able to demonstrate a significant reduction in the incontinence symptoms in the subjects the investigators asses that vibration can be a way of reestablishing a normal function of the pelvic floor muscles and bladder function in incontinent patients.

ELIGIBILITY:
Inclusion Criteria:

* Women suffering from stress incontinence OR Women suffering from urge incontinence /overactive bladder syndrome
* Ongoing anticholinergic treatment in the urge incontinence/overactive bladder syndrome group
* Patient capable of understanding protocol and performing treatment

Exclusion Criteria:

* On going pregnancy or breast feeding
* Treatment with anticholinergic medications in the stress incontinence group
* Treatment with diuretic drugs
* Acute illness (including infection, trauma and haematuria)
* Fibromyalgia
* Faecal incontinence
* Known neurological disease
* Bladder pain syndrome
* Genital prolaps > stage 2 on the Pelvic Organ Prolapse Quantification System POP-Q
* Previous treatment with neuromodulation or Botox
* Previous pelvic floor surgery or radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Diaper test - weight (grams) | Assesment at baseline and again after 6 weeks of treatment (when treatment is terminated)

SECONDARY OUTCOMES:
Validated symptom score (ICI-Q) including: changes in incontinence and micturition patterns; patients' subjective assessment of their symptoms | Assesment at baseline and again after 6 weeks of treatment (when treatment is terminated)
Treatment satisfaction | After 6 weeks of treatment (when treatment is terminated)
Urethral pressure (in the stress group) | Assesment at baseline and again after 6 weeks of treatment (when treatment is terminated)
Episodes of over active bladder during urodynamics (urge patients) | Assesment at baseline and again after 6 weeks of treatment (when treatment is terminated)
Micturition diary - The number of involuntary incontinence and normal micturition episodes | Assesment at baseline and again after 6 weeks of treatment (when treatment is terminated)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Fode, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Departement of Gynecology, Roskilde Hospital, Roskilde, Denmark, Denmark